CLINICAL TRIAL: NCT02919891
Title: The Relationship of Intra-epidermal Nerve Fibre Density (IENFD) and Structure to Chronic Post-Mastectomy Pain Syndrome (PMPS)
Brief Title: Relationship of Intra-Epidermal Nerve Fibre Density (IENFD) and Structure to Chronic Post-Mastectomy Pain Syndrome (PMPS)
Status: Completed | Type: Observational
Sponsor: Royal Infirmary of Edinburgh (Other)
Responsible Party: Principal Investigator, Oliver Daly, Consultant Anaesthetist, Royal Infirmary of Edinburgh
Other Study IDs: R&D no. 2016/0081
Record Dates: First submitted 2016-08-25; First posted 2016-09-29 (Estimated); Last update posted 2018-04-11 (Actual); Status verified 2018-04

CONDITIONS: Chronic Pain; Pain Measurement; Mastectomy; Postoperative Pain
Keywords: intra-epidermal nerve fibre density; IENFD; Chronic Pain; Post-mastectomy; Post-mastectomy pain syndrome; PMPS; Chronic Post-Surgical Pain; CPSP; Mastectomy
MeSH Terms: conditions — Chronic Pain; Pain, Postoperative | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Participants with Chronic Pain: Questionnaire results will allow the diagnosis of chronic pain. No intervention will be administered. The results of the IENFD will be compared to the group without chronic pain.
  Interventions: Other: Questionnaire
- Participants without Chronic Pain: Questionnaire results will reveal the absence of chronic pain. No intervention will be administered. The results of the IENFD will be compared to the group with chronic pain.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Questionnaires

SUMMARY:
This is a retrospective, observational study which will utilise the Edinburgh Cancer Research Centre's Tissue Bank to provide samples for IENFD testing in those who have undergone mastectomy surgery for breast cancer.

The investigators shall identify all those patients in the Tissue Bank database who have undergone mastectomy surgery for breast cancer. The investigators shall consult the patient's electronic health record, and general practitioner if required, to ascertain whether the patient has died, been diagnosed with cognitive impairment or a psychotic disorder, or receiving ongoing oncological treatment which would exclude them from the study. The investigators shall also exclude all those patients who received surgery within the last year as we intend to elucidate the presence of pain in the immediate post-operartive period up to 12 months post-operatively.

Having identified these patients the investigators shall contact them via post with a pack containing an information document, a consent form and questionnaires. As this is an observational study we shall contact all of the identified patients who meet the inclusion criteria with the aim of recruiting as many as possible. The investigators would anticipate a high response rate as has been the experience with previous questionnaire studies of breast cancer patients.

Once a signed consent form has been returned the patient's tissue sample would undergo IENFD testing. Their questionnaire responses will allow participants to be split into two groups based upon whether they experience CPSP or not. Blinding of this grouping will take place so that those undertaking the IENFD testing are unaware of the patient's questionnaire responses.

Statistical analysis of the two group's IEFD results and questionnaire responses will then be undertaken with the null hypothesis that the pre-operative IENFD at the site of surgery does not predict or correlate with CPSP.

DETAILED DESCRIPTION:
Study Design This study will use pre-existing skin samples stored in the Edinburgh Experimental Cancer Medicine Centre (ECMC) / SAHSC BioResource (collected from 2006-2012) from patients who have undergone breast cancer surgery.

The investigators shall firstly identify all samples in the Tissue Bank database that were taken from those undergoing breast cancer surgery. Before any patient details are provided the investigators will confirm that the patient has initialled the following section of the consent form they completed at the time of their surgery;

"I agree to my name and details being made available to other ECMC researchers who might approach me to invite participation in other research projects. These might include studies of new treatments or techniques, clinical or genetic studies of the causes of cancer or cancer outcomes. I understand that that this permission does not commit me to participate in such studies and I will be able to decide whether I wish to be involved once I have reviewed any information sheet and consent form."

Once this has been confirmed, the investigators shall consult the patient's electronic health record to ascertain whether anything would exclude them from the study such as death, a new diagnosis of cognitive impairment or a psychotic disorder, or receiving current oncological treatment.

As this is an exploratory study the investigators shall contact all of the identified patients who meet the inclusion criteria with the aim of recruiting as many as possible. The investigators would anticipate a high response rate, as has been the experience with previous questionnaire studies involving breast cancer patients.

The investigators will contact the identified patients via post with a pack containing a cover letter from the principal investigator of the original clinical team, an information document, a consent form and questionnaires. The information document will include contact details of the principal investigator and research team to allow patients to discuss the study, ask questions that they have, or ask for assistance from the research team in any aspect of completing the documentation. The questionnaires are the only requirement of participants to complete for the study and should take less than 30 minutes to do so. The questionnaires include the Hospital Anxiety and Depression Score (HADS), the EQ-5D, the Brief Pain Inventory (BPI), the Short-form McGill Pain Questionnaire-2 and the Short Leeds Assessment of Neuropathic Symptoms and Signs (S-LANSS) which are all commonly used scoring tools for chronic pain. There is no need for a hospital visit, physical examination,or blood tests.

After 4-6 weeks, if no response is received from an individual patient we would send a second letter to ensure that the initial pack had been received.

Once a signed consent form and questionnaires have been returned, a paper Case Report Form (CRF) will be created with a unique study number which will be added to the questionnaires as the only identifying information. The unique number currently given to the Edinburgh Experimental Cancer Medicine Centre (ECMC) / SAHSC BioResource samples held for the patient will also be added to the CRF. In this way, both those carrying out the laboratory work and the questionnaire data entry will only be provided with an identifying number and be blinded since they have no access to the CRF.

The Edinburgh Experimental Cancer Medicine Centre (ECMC) / SAHSC BioResource samples shall be serially cut with a microtome to produce 8 micron thick sections with three sections per sample created to ensure consistency. The sections shall then be stained with neurofilament and anti-protein gene product (anti-PGP) 9.5 and examined under bright field microscopy. An image of the section shall be captured and analysed by the same individual using Image J software to calculate the IENFD.

Once all samples have been analysed the CRF would be used to place the IENFD results into two groups based upon their questionnaire responses. These two groups would be those with and those without CPSP symptoms.

Statistical analysis of the two group's IEFD results and questionnaire responses will then be undertaken with the null hypothesis that the pre-operative IENFD at the site of surgery does not predict or correlate with CPSP.

Study Centres Recruitment of all patients will take place from the Edinburgh Cancer Research Centre (ECRC) at the Western General Hospital.

Timelines and Consent The investigators would expect that reading the cover letter and information pack, signing the consent form, and completing the questionnaires will take between 20 and 30 minutes. The investigators aim to recruit patients over a 3 - 6 month period before moving on to performing IENFD testing over the next 6 - 9 months. A further 3 - 6 months will be required to analyse and present our results.

The patients have already consented for their tissue sample to be used in future research. Consent will be sought for the patient to complete the questionnaires which are essential to the study in order to identify those who have developed CPSP.

There is no ongoing intervention or follow-up for the patients themselves after they consent to inclusion in the study. However, if in completing the questionnaire they become aware of suffering from CPSP we provide details of how to be referred to a pain specialist if they feel it would be of benefit. To facilitate this we would contact their general practitioner with details of how to refer a patient such as via the SCI Gateway Advice Service or Lothian Chronic Pain Service Email Advice Service.

ELIGIBILITY:
Inclusion Criteria:

* Patient has Tissue Bank sample stored in the Edinburgh Experimental Cancer Medicine Centre (ECMC) / SAHSC BioResource.
* At the time of their surgery, the patient provided written consent for the sample to be used by future researchers and to be contacted by those researchers.
* Patient has undergone surgery for breast cancer.
* Contact details for the patient are available.
* Patient is able to provide informed consent for the questionnaire component of the study.
* Patient is able to complete and return study questionnaires. Telephone support to help complete the study documentation will be provided if requested.

Exclusion Criteria:

* Patient who had their surgery outwith the timeframe of the original study consent (2006-2012)
* Patients receiving active oncological treatment.
* Patients who have died.
* Patients with cognitive impairment or significant mental health disorder.
* Patients with active complications of their surgical wound site.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients that have undergone mastectomy surgery with a Tissue Bank sample stored in the Edinburgh Experimental Cancer Medicine Centre (ECMC) / SAHSC BioResource.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
Relationship of intra-epidermal nerve fibre density to the presence of post-mastectomy pain syndrome as assessed by validated questionnaires | From time of original surgery to current date - could be up to 5 years after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Oliver Daly, Edinburgh, Midlothian, United Kingdom

IPD SHARING:
Plan to Share IPD: No